CLINICAL TRIAL: NCT03811457
Title: Immunotherapy With CD19 CAR T-cells in Patients With Relapsed or Refractory CD19+ Leukemia and Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UWELL Biopharma (Industry)
Collaborators: Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCAR019
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Lymphoma Leukemia
Keywords: CAR-T cell, CD19, Lymphoma, Leukemia
MeSH Terms: conditions — Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Welgenaleucel (UWC19) (Experimental): The Chimeric Antigen Receptor T Cell Immunotherapy (CAR-T) Dosage form：injection Dosage: 100mL in total Frequency:the first day, the second day, the third day Duration:total three times
  Interventions: Genetic: Welgenaleucel

INTERVENTIONS:
Genetic: Welgenaleucel — Welgenaleucel (UWC19) is a CD19-directed immunotherapy consisting of autologous T cells, which is reprogrammed to target cells that express CD19.
  Other Names: UWC19

SUMMARY:
B cell malignancies comprise a heterogeneous group of neoplasms including a vast majority of non-Hodgkin's lymphomas (NHL), lymphoblastic leukemias (ALL) and chronic lymphocytic leukemias (CLL). Current treatments for B cell malignancies include chemotherapy, radiation therapy, bone marrow transplantation, and peripheral blood stem cell transplantation. Despite these treatment modalities, most patients will remain incurable. Welgenaleucel (UWC19) is a CD19-directed genetically-modified autologous immunotherapy. This study is designed to evaluate safety and feasibility of administering Welgenaleucel (UWC19) transduced with anti-CD19 lentiviral vector to patients with advanced refractory hematologic malignancies, including DLBCL and ALL.

ELIGIBILITY:
Inclusion Criteria:

* CD19+ leukemia or lymphoma patients with no available curative treatment options who have limited prognosis with currently available therapies
* Absolute lymphocyte count, ALC )≧600/μl
* HIV, HTLV, Syphilis negative
* GPT ≦200 U/L
* Cr ≦221 umol/L
* Adequate venous access for apheresis, and no other contraindications for leukapheresis.
* Voluntary informed consent is given.

Exclusion Criteria:

* Body weight < 20Kg
* Pregnant women.
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection.
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
* Previously treatment with any gene or cell therapy products.
* Any uncontrolled active medical disorder that would preclude participation as outlined.
* Expected survival< 12 weeks
* Received investigational drug or device within 30 days pre-trial;
* Patients with any other serious diseases considered by the investigator(s) not in the condition to enter the trial.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The adverse events associated with CAR T cell product infusions are assessed. | 30 days
  The type, frequency, severity, and duration of adverse events will be summarized

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Yi Kuo, PhD, Study Director — UWELL Biopharma
Locations (1):
- Liaocheng People Hospital, Liaocheng, Shandong, China